CLINICAL TRIAL: NCT01590069
Title: Phase I/II Study of Aerosol Interleukin-2 for Pulmonary Metastases
Brief Title: Aerosolized Aldesleukin in Treating Patients With Lung Metastases
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0700; NCI-2012-00788 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0700; 2010-0700 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Malignant Neoplasm in the Lung; Metastatic Melanoma; Metastatic Osteosarcoma; Metastatic Renal Cell Cancer; Sarcoma; Stage IV Cutaneous Melanoma AJCC v6 and v7; Stage IV Osteosarcoma AJCC v7; Stage IV Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Melanoma; Osteosarcoma; Carcinoma, Renal Cell; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (aerosolized aldesleukin) (Experimental): Patients receive aerosolized aldesleukin QD on days 1-21. Courses repeat every 28 days in the absence of disease progression of unacceptable toxicity.
  Interventions: Biological: Aerosolized Aldesleukin; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Aerosolized Aldesleukin — Breathe aerosolized aldesleukin
  Other Names: Aerosolized Recombinant IL-2
Other: Laboratory Biomarker Analysis — Optional correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of aerosolized aldesleukin and to see how well it works in treating patients with cancer that has spread from the original tumor to the lungs. Biological therapies, such as aerosolized aldesleukin, may stimulate or suppress the immune system in different ways and stop tumor cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate toxicity in patients with lung metastases during aerosol interleukin (IL)-2 (aldesleukin) therapy using self-report, remote spirometry and pulse oximetry.

SECONDARY OBJECTIVES:

I. To determine dose and schedule of an acceptable aerosol IL-2 regimen and correlate with absolute lymphocyte count (ALC).

II. To determine serum IL-2 levels on day 1 of therapy for evidence of spillover into circulation and correlate with absence or presence of toxicity.

III. To evaluate the efficacy of aerosol IL-2 treatment using Response Evaluation Criteria in Solid Tumors (RECIST).

TERTIARY OBJECTIVES:

I. To evaluate the histology in post-surgical specimens in patients who undergo surgery for lung metastases following aerosol IL-2 treatment as an optional procedure.

II. To evaluate immune correlates from optional pre-treatment biopsy and post-surgical specimen.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive aerosolized aldesleukin once daily (QD) on days 1-21. Courses repeat every 28 days in the absence of disease progression of unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of advanced cancer with lung metastases; patients with no prior therapy are eligible if there is no known superior alternative medical therapy; for phase Ib expansion cohort diagnosis of osteosarcoma, lung metastases will be required
* Willing to comply with protocol therapy and required safety monitoring (self-report, pulse oximetry, remote spirometry, labs)
* Creatinine =< 2 x upper limit of normal (ULN)
* Bilirubin =< 5 x ULN
* Aspartate aminotransferase (AST) =< 5 x ULN
* Forced vital capacity (FVC) >= 50% predicted
* Oxygen (O2) saturation at rest >= 90% (off supplementary oxygen)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 for ages >= 16 or Lansky play >= 80% for ages =< 15
* Patients must have recovered to =< grade 1 toxicity (except alopecia and hearing loss) from any prior chemotherapy, other investigational therapy, hormonal, biological, targeted agents
* No radiotherapy within 2 weeks: exception: patients may receive palliative low dose radiotherapy (30 Gy or less) for lesions outside the lung at the discretion of the treating physician; palliative radiotherapy could be given before aerosol treatment is started if necessary
* Subjects have to be able to read and understand English
* Patients with advanced cancer with resectable lung metastases
* Patients with sarcoma, renal cell carcinoma, or melanoma or with known disease outside the lungs and/or thorax

Exclusion Criteria:

* Currently being treated with bronchodilators or corticosteroids
* Females: pregnant or breast feeding and if of child bearing potential (e.g. female of childbearing age that has not been amenorrheic for at least 12 consecutive month or surgically sterilized) not willing to use effective contraception
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, bradycardia, related to cardiac disease, bundle branch block, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Subjects with baseline symptoms of fever and/or cough and/or shortness of breath and/or wheezing and/or fatigue grade >= 2 (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 4.0)
* Patients with unresectable lung metastases
* Patients without sarcoma, renal cell carcinoma, or melanoma

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-06-28 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose, defined as the highest dose level with six patients with at most one dose limiting toxicity, using the CTCAE v4.0 (Phase I) | 28 days
  The dose escalation will be conducted via the accelerated titration method for the first 2 dose levels.
Incidence of adverse events (AE)s, using the CTCAE v4.0 (Phase II) | Up to 4 years
  AEs will be summarized by severity according to the worst grade experienced over the number of patients at risk.
Response of measurable lesions to aerosol aldesleukin using modified RECIST (Phase II) | Up to 4 years
  Response analysis will be performed on intent-to-treat, that is, any patient who enrolled into the expansion cohort. Patients who withdraw before the end of 2 months without responding will be considered non-responders. The two-sided 95% Clopper-Pearson confidence intervals will be calculated for the proportion of patients with responses.

SECONDARY OUTCOMES:
IL-2 levels in serum | Day 1 of therapy
  Serum IL-2 levels will be compared with maximum grade of toxicity to determine whether our hypothesis of "spillover" of IL-2 in the circulation - i.e. some escaping the receptor gauntlet of IL-2 receptor bearing cells in pulmonary lymphatics.
Changes in biomarker levels | Baseline to 8 weeks
  Changes in biomarker levels between pre- and post-treatment tissue samples will be assessed using paired t-tests (if the data are normally distributed) or Wilcoxon signed-rank tests (otherwise). Will graph the data using histograms, box plots and dot plots. With 20 patients, using a 2-sided 5% alpha, there would be 80% power to detect an effect size of 0.66 (where the effect size is the mean difference divided by the standard deviation of the differences).

CONTACTS AND LOCATIONS:
Overall Officials: Najat Daw, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org